CLINICAL TRIAL: NCT01538836
Title: Calorie Restriction and Metabolic Health
Brief Title: Calorie Restriction, Protein Supplementation and Metabolic Health
Acronym: CRPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRPS-201107354; 1R01DK094483-01A1 (NIH)
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Obesity; Menopause; Osteoporosis; Sarcopenia
MeSH Terms: conditions — Obesity; Osteoporosis; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Weight maintenance (No Intervention): Weight maintenance with normal protein intake
- Weight loss with normal protein intake (Active Comparator)
  Interventions: Behavioral: Weight loss with normal protein intake
- Weight loss with protein supplementation (Experimental)
  Interventions: Behavioral: Weight loss with protein supplementation

INTERVENTIONS:
Behavioral: Weight loss with normal protein intake — Goal of 8 to 10% weight loss while consuming the recommended daily allowance of protein (i.e, 0.8 grams of protein per kg body weight per day).
  Arms: Weight loss with normal protein intake
Behavioral: Weight loss with protein supplementation — Goal of 8 to 10% weight loss while consuming 150% of the recommended daily allowance of protein (i.e., 1.2 grams of protein per kg body weight per day).
  Arms: Weight loss with protein supplementation

SUMMARY:
The purpose of this study is to determine whether consuming additional protein during calorie restriction induced weight loss has beneficial or harmful effects on multi-organ (liver, muscle, adipose tissue) insulin sensitivity, colonocyte proliferation rates, the gut microbiome, muscle mass and function, and bone mineral density in obese, postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Obese with body mass index (BMI) between 30 and 50 kg/m2
* Postmenopausal
* Sedentary (i.e., less than 1.5 hours of exercise per week)

Exclusion Criteria:

* Individuals with diabetes and/or uncontrolled hypertension
* Individuals with hepatitis B and/or C
* Individuals who smoke
* Individuals with an allergy to whey protein

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in muscle volume | Baseline and at 10% weight loss in calorie restriction groups and ~6 to 7 months in the weight maintenance group
  Thigh muscle volume will be measured by magnetic resonance imaging (MRI)
Change in muscle strength | Baseline and at 10% weight loss in calorie restriction groups and ~6 to 7 months in the weight maintenance group
  Muscle strength will be evaluated by administering maximum one repetition strength and isokinetic strength tests.
Changes in bone mineral density and bone mineral content | Baseline and at 10% weight loss in calorie restriction groups and ~6 to 7 months in the weight maintenance group
  Total bone mass and total body and regional bone mineral density will be evaluated by using dual X-ray energy absorptiometry (DXA).

SECONDARY OUTCOMES:
Change in insulin sensitivity | Baseline and at 10% weight loss in calorie restriction groups and ~6 to 7 months in the weight maintenance group
  Insulin sensitivity (glucose rate of disappearance [Rd] during a hyperinsulinemic-euglycemic clamp procedure) will be evaluated in a subset of 10 participants per group because power analysis has determined that this number is sufficient to detect a 25% difference between groups assuming 80% power, an alpha value of 0.05 and an average baseline insulin-stimulated glucose Rd of 2,590 ± 492 µmol/min, the average ± SD insulin stimulated glucose Rd the investigators have measured during the past 20 y in obese subjects. In the investigators' experience (Kirk et al., 2009 and Magkos et al., 2016), the weight loss induced increase in insulin stimulated glucose Rd is ~50%.
Change in muscle protein metabolism | Baseline and at 5% weight loss in the calorie restriction groups and after ~3 months in the weight maintenance group
  Rates of muscle protein synthesis, breakdown and net protein balance will be assessed during postabsorptive conditions and when insulin and/or amino acid concentrations are elevated.
Change in bacterial populations found in the stool | Baseline and at 10% weight loss in calorie restriction groups and ~6 to 7 months in the weight maintenance group
Change in cell proliferation (growth) rates in the colon | Baseline and at 10% weight loss in calorie restriction groups and ~6 to 7 months in the weight maintenance group
  Colon cell proliferation rates will be determined using stable isotope labelled tracer methods in conjunction with sigmoid colon biopsy samples
Determine the acute effect of whey protein ingestion on skeletal muscle insulin sensitivity | Prior to starting the weight loss or maintenance intervention
  Insulin sensitivity will be evaluated using the hyperinsulinemic-euglycemic clamp procedure in conjunction with stable isotope labeled tracer infusions
Determine the acute effect of whey protein ingestion on muscle protein metabolism | Prior to starting the weight loss or maintenance intervention
  Rates of muscle protein synthesis, breakdown and net protein balance will be assessed using stable isotope labeled tracer methods during postabsorptive conditions and during insulin infusion with or without whey protein ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Mittendorfer, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Kirk E, Reeds DN, Finck BN, Mayurranjan SM, Patterson BW, Klein S. Dietary fat and carbohydrates differentially alter insulin sensitivity during caloric restriction. Gastroenterology. 2009 May;136(5):1552-60. doi: 10.1053/j.gastro.2009.01.048. Epub 2009 Jan 25. PMID 19208352
- [Background] Magkos F, Bradley D, Eagon JC, Patterson BW, Klein S. Effect of Roux-en-Y gastric bypass and laparoscopic adjustable gastric banding on gastrointestinal metabolism of ingested glucose. Am J Clin Nutr. 2016 Jan;103(1):61-5. doi: 10.3945/ajcn.115.116111. Epub 2015 Nov 25. PMID 26607940
- [Result] Smith GI, Yoshino J, Kelly SC, Reeds DN, Okunade A, Patterson BW, Klein S, Mittendorfer B. High-Protein Intake during Weight Loss Therapy Eliminates the Weight-Loss-Induced Improvement in Insulin Action in Obese Postmenopausal Women. Cell Rep. 2016 Oct 11;17(3):849-861. doi: 10.1016/j.celrep.2016.09.047. PMID 27732859
- [Result] Smith GI, Patterson BW, Klein SJ, Mittendorfer B. Effect of hyperinsulinaemia-hyperaminoacidaemia on leg muscle protein synthesis and breakdown: reassessment of the two-pool arterio-venous balance model. J Physiol. 2015 Sep 15;593(18):4245-57. doi: 10.1113/JP270774. Epub 2015 Aug 14. PMID 26150260
- [Result] Smith GI, Yoshino J, Stromsdorfer KL, Klein SJ, Magkos F, Reeds DN, Klein S, Mittendorfer B. Protein Ingestion Induces Muscle Insulin Resistance Independent of Leucine-Mediated mTOR Activation. Diabetes. 2015 May;64(5):1555-63. doi: 10.2337/db14-1279. Epub 2014 Dec 4. PMID 25475435
- [Derived] Smith GI, Commean PK, Reeds DN, Klein S, Mittendorfer B. Effect of Protein Supplementation During Diet-Induced Weight Loss on Muscle Mass and Strength: A Randomized Controlled Study. Obesity (Silver Spring). 2018 May;26(5):854-861. doi: 10.1002/oby.22169. PMID 29687650
- [Derived] Harris LLS, Smith GI, Patterson BW, Ramaswamy RS, Okunade AL, Kelly SC, Porter LC, Klein S, Yoshino J, Mittendorfer B. Alterations in 3-Hydroxyisobutyrate and FGF21 Metabolism Are Associated With Protein Ingestion-Induced Insulin Resistance. Diabetes. 2017 Jul;66(7):1871-1878. doi: 10.2337/db16-1475. Epub 2017 May 4. PMID 28473464